CLINICAL TRIAL: NCT01205451
Title: A Multicenter, Open-label, Single Dose Study of the Safety and Efficacy of GSK1358820 (Botulinum Toxin Type A) in Chinese Subjects With Post-stroke Focal Upper Limb Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114609
Record Dates: First submitted 2010-09-03; First posted 2010-09-20 (Estimated); Results first posted 2012-09-24 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Spasticity, Post-Stroke
Keywords: GSK1358820; upper limb; spasticity; post-stroke
MeSH Terms: conditions — Muscle Spasticity | interventions — Botulinum Toxins, Type A

ARMS (1):
- BTX-A (Experimental): Botulinum toxin type A
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin type A

SUMMARY:
This trial is a multicenter, open-label study to evaluate the safety and efficacy of GSK1358820 for treatment in post-stroke subjects with focal wrist, finger and in some cases, thumb spasticity. Qualified patients who complete GSK double-blind study 112958 will be enrolled. Subjects will receive a single treatment session of intramuscular GSK1358820 "200U or 240U (if thumb spasticity is present)". The subjects will be observed until 12 weeks post injection. Outcome measures include changes from baseline at every post injection visit as measured on the Modified Ashworth Scale (MAS), Disability Assessment Scale (DAS) and Global Assessment Scale. Safety parameters will be measured including adverse events, vital signs (pulse and blood pressure) and clinical laboratory tests (haematology, serum chemistry and urinanalysis).

DETAILED DESCRIPTION:
This trial is a multicenter, open-label study to evaluate the safety and efficacy of GSK1358820 for the treatment of patients with focal wrist, finger and in some cases, thumb spasticity post-stroke. Qualified patients will be eligible for enrollment upon completion of double-blind study 112958. Patients will receive a single treatment session with intramuscular injections of GSK1358820 "200U or 240U (if thumb spasticity is present)".The subjects will be observed for 12 weeks post injection.

Each completed subject will attend 4 clinic visits. The maximum study duration is 13 weeks. The study includes a 1 week pretreatment period, during which the screening visit (visit 1 could be the last visit of previous double-blind study 112958 or any time within 3 months after completion of previous study) is to take place. Only one upper limb (meeting inclusion/exclusion criteria) will be evaluated and treated in the study. Subjects will receive a single intramuscular treatment with investigated drug at day 0 (visit 2). There will be two post-injection follow-up visits at week 6 and 12 (visits 3 to 4).

ELIGIBILITY:
Inclusion Criteria:

1. Within 3 months after completion of the GSK/Allergan study 112958.
2. Wrist flexor muscle tone of 2 or greater and finger flexor muscle tone of 1 or greater as measured on MAS (0 to 4).
3. At least one functional disability item (i.e., hygiene, dressing, pain, or cosmesis) with a rating of 2 or greater on DAS (0 to 3).
4. If using physical therapy, must be stable for at least 1 month prior to study enrolment in study 112958.
5. >=40kg in weight.
6. QTc criteria: (either QTcb or QTcf, machine or manual overread, males or females); include the following details as appropriate: QTc<450 millisecond (msec) or <480msec for subjects with Bundle Branch Block - values based on either single electrocardiogram (ECG) values or triplicate ECG averaged QTc values obtained over a brief recording period.
7. Liver function tests: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2xULN; alkaline phosphatase and bilirubin ≤1.5xULN (isolated bilirubin >1.5ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
8. In the opinion of the investigator, subject must clearly understand the intent of the study and be willing and able to comply with study instructions and complete the entire study.
9. Informed consent has been obtained

Exclusion Criteria:

1. Presence of fixed contracture of the study limb (absence of passive range of motion).
2. Profound atrophy of muscles to be injected (in the investigators opinion).
3. Infection or dermatological condition at the injection sites.
4. Significant inflammation in the study limb limiting joint movement.
5. History of or planned treatment for spasticity with phenol or alcohol block in the study limb.
6. History of or planned surgical intervention for spasticity of the study limb.
7. History (within 3 months of qualification) of or planned (during study period) casting of the study limb.
8. Participation in another clinical study (with the exception of study 112958) , within the 30 days immediately prior to enrolment.
9. Planned or anticipated initiation of new antispasticity medications during the clinical study.
10. Any medical condition that may put the subject at increased risk with exposure to GSK1358820, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other disorder that might have interfered with neuromuscular function.
11. Concurrent use of aminoglycoside antibiotics or other agents that might interfere with neuromuscular function. A full list of prohibited medications that interfere with neuromuscular transmission is provided as Appendix 1.
12. Current treatment for spasticity with an intrathecal baclofen.
13. Females who are pregnant, nursing, or planning a pregnancy during the study period, or females of childbearing potential, not using a reliable means of contraception.
14. Known allergy or sensitivity to study medication or its components.
15. Bedridden subjects.
16. Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
17. Presence of clinically unstable severe cardiovascular, renal or respiratory disease.
18. Investigator's opinion that the subject has a concurrent condition(s) that may put the subject at significant risk, may confound the study results, or may interfere significantly with the conduct of the study.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- China (10):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Haerbin, Heilongjiang
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Suzhou, Jiangsu
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Shanghai

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study LOC114609 (NCT01205451) is the open-label (OL) extension of Study 112958 (a double-blind [DB] study; NCT01153815). Within 3 months of completion of Study 112958, eligible participants were enrolled in Study 114609.
Groups:
- BOTOX in Original DB Study; BOTOX in OL Study: Participants who had received Botulinum Toxin Type A (BOTOX or GSK1358820) treatment in the previous double-blind study (Study 112958) received BOTOX 200 Units (U) (4 milliliters [mL]) injected into the wrist and finger muscles in this open-label extension study. 40 U (0.8 mL) was injected into the thumb muscles if thumb spasticity was present during the 12-week study (once at Week 0).
- Placebo in Original DB Study; BOTOX in OL Study: Participants who had received placebo treatment in the previous double-blind study (Study 112958) received BOTOX 200 Units (U) (4 milliliters [mL]) injected into the wrist and finger muscles in this open-label extension study. 40 U (0.8 mL) was injected into the thumb muscles if thumb spasticity was present during the 12-week study (once at Week 0).
Period: Overall Study
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Started | 53 | 56
Completed | 47 | 46
Not Completed | 6 | 10
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics are summarized for members of the Full Analysis Set (FAS), comprised of all enrolled and treated participants with at least one post-treatment modified Ashworth scale (MAS) wrist score. Three participants (all receiving placebo in the original DB study) didn't have any post-treatment MAS wrist score; therefore, the FAS included 106 participants (53 participants in each group).
  Years | 54.4 (10.90) | 55.4 (12.53) | 54.9 (11.70)
Gender [Count of Participants; unit: Participants] — Baseline characteristics are summarized for members of the Full Analysis Set (FAS), comprised of all enrolled and treated participants with at least one post-treatment MAS wrist score. Three participants (all receiving placebo in the original DB study) didn't have any post-treatment MAS wrist score; therefore, the FAS included 106 participants (53 participants in each group).
  Participants
    Female | 10 | 10 | 20
    Male | 43 | 43 | 86
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics are summarized for members of the Full Analysis Set (FAS), comprised of all enrolled and treated participants with at least one post-treatment MAS wrist score. Three participants (all receiving placebo in the original DB study) didn't have any post-treatment MAS wrist score; therefore, the FAS included 106 participants (53 participants in each group).
  participants
    Chinese | 53 | 53 | 106
Number of participants with the absence or presence of thumb spasticity [Number; unit: participants] — Baseline characteristics are summarized for members of the Full Analysis Set (FAS), comprised of all enrolled and treated participants with at least one post-treatment MAS wrist score. Three participants (all receiving placebo in the original DB study) didn't have any post-treatment MAS wrist score; therefore, the FAS included 106 participants (53 participants in each group).
  participants
    Absence | 6 | 6 | 12
    Presence | 47 | 47 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 6 and Week 12 for Wrist Flexor Muscle Tone as Measured on the Modified Ashworth Scale (MAS)
Description: The investigator or assessor extended the participant's wrist as quickly as possible to grade flexor muscle tone. The MAS wrist score was calculated by using the 6-point MAS (0, 1, 1+ [regarded as 1.5], 2, 3, and 4; 0=no increase in muscle tone; 4=affected part[s] rigid in flexion/extension). Change from Baseline at Week 6 or Week 12 was calculated as the value at Week 6 or Week 12 minus the value at Baseline.
Time Frame: Baseline (Day 0), Week 6, and Week 12
Population: Full Analysis Set (FAS) Population: all randomized and treated participants with at least one post-treatment MAS wrist score. The missing data imputation method was used for analysis. For each participant, missing data points were replaced by the mean of the non-missing scores from both treatment groups for that variable at the specific visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 53 | 53
scores on a scale
  Week 6 | -1.21 (0.616) | -1.33 (0.753)
  Week 12 | -0.88 (0.589) | -1.12 (0.752)
Statistical Analysis 1: Comparison: BOTOX in Original DB Study; BOTOX in OL Study; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — The P-value for change from Baseline indicates the comparision of the Week 6 value against the Baseline value; t-distribution = -1.21, 95% CI 2-sided [-1.38 to -1.04] — Confidence intervals for means were based on the t-distribution
Statistical Analysis 2: Comparison: Placebo in Original DB Study; BOTOX in OL Study; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — The P-value for change from Baseline indicates the comparision of the Week 6 value against the Baseline value; t-distribution = -1.33, 95% CI 2-sided [-1.54 to -1.12] — Confidence intervals for means were based on the t-distribution
Statistical Analysis 3: Comparison: BOTOX in Original DB Study; BOTOX in OL Study; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — The P-value for change from Baseline indicates the comparision of the Week 12 value against the Baseline value; t-distribution = -0.88, 95% CI 2-sided [-1.04 to -0.72] — Confidence intervals for means were based on the t-distribution
Statistical Analysis 4: Comparison: Placebo in Original DB Study; BOTOX in OL Study; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — The P-value for change from Baseline indicates the comparision of the Week 12 value against the Baseline value; t-distribution = -1.12, 95% CI 2-sided [-1.33 to -0.91] — Confidence intervals for means were based on the t-distribution

2. Secondary Outcome: Number of Participants Classified as Wrist Treatment Responders at Week 6 and Week 12
Description: Wrist treatment responders are defined as participants with a decrease in wrist flexor muscle tone of at least one point on the MAS from Baseline. The MAS wrist score was calculated by using the 6-point MAS (0, 1, 1+ [regarded as 1.5], 2, 3, and 4; 0=no increase in muscle tone; 4=affected part[s] rigid in flexion/extension).
Time Frame: Baseline (Day 0), Week 6, and Week 12
Population: FAS Population. The missing data imputation method was used for analysis.
Measure: Number; unit: participants
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 53 | 53
participants
  Week 6 | 43 | 42
  Week 12 | 35 | 39

3. Secondary Outcome: Change From Baseline at Week 6 and Week 12 for Finger Flexor Muscle Tone as Measured on the MAS
Description: The investigator or assessor extended the participant's finger as quickly as possible to grade the flexor muscle tone. The MAS finger score was calculated by using the 6-point MAS (0, 1, 1+ [regarded as 1.5], 2, 3, and 4; 0=no increase in muscle tone; 4=affected part[s] rigid in flexion/extension). Change from Baseline at Week 6 or Week 12 was calculated as the value at Week 6 or Week 12 minus the value at Baseline.
Time Frame: Baseline (Day 0), Week 6, and Week 12
Population: FAS Population. The missing data imputation method was used for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 53 | 53
scores on a scale
  Week 6 | -1.14 (0.716) | -1.29 (0.769)
  Week 12 | -0.72 (0.607) | -0.96 (0.805)

4. Secondary Outcome: Change From Baseline at Week 6 and Week 12 for Thumb Flexor Muscle Tone as Measured on the MAS
Description: The investigator or assessor extended the participant's thumb as quickly as possible to grade the flexor muscle tone. The MAS thumb score was calculated by using the 6-point MAS (0, 1, 1+ [regarded as 1.5], 2, 3, and 4; 0=no increase in muscle tone; 4=affected part[s] rigid in flexion/extension). Change from Baseline at Week 6 or Week 12 was calculated as the value at Week 6 or Week 12 minus the value at Baseline.
Time Frame: Baseline (Day 0), Week 6, and Week 12
Population: FAS Population. Only those participants who had thumb spasticity were analyzed. The missing data imputation method was used for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 47 | 47
scores on a scale
  Week 6 | -1.02 (0.642) | -1.22 (0.721)
  Week 12 | -0.80 (0.631) | -0.92 (0.716)

5. Secondary Outcome: Change From Baseline at Week 6 and Week 12 for the Principal Measure as Assessed on the Disability Assessment Scale (DAS)
Description: The investigator assessed 4 areas of disability, hygiene, pain, dressing, and limb posture, using the 4-point DAS (0=No functional disability to 3=Severe disability). Prior to the first dose, the investigator, in consultation with the participant, selected 1functional disability item (which had to have a score of 2 or greater as measured on the DAS, indicating moderate to severe disability) from the 4 areas of disability and assessed it as a principal measure. Change from Baseline at Week 6 or Week 12 was calculated as the value at Week 6 or Week 12 minus the value at Baseline.
Time Frame: Baseline (Day 0), Week 6, and Week 12
Population: FAS Population. The missing data imputation method was used for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 53 | 53
scores on a scale
  Week 6 | -0.64 (0.591) | -0.72 (0.662)
  Week 12 | -0.59 (0.570) | -0.57 (0.665)

6. Secondary Outcome: Global Assessment Scale (GAS) Score as Evaluated by the Physician at Week 6 and Week 12
Description: The physician used the GAS to assess response to treatment at each visit after injection. The assessor was the same throughout the study period. GAS scores were assessed by using the 9-point GAS (-4, -3, -2, -1, -0, +1, +2, +3, +4; -4=very marked worsening, -0=unchanged, +4=very marked improvement) at Week 6 and Week 12.
Time Frame: Week 6 and Week 12
Population: FAS Population. The missing data imputation method was used for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 53 | 53
scores on a scale
  Week 6 | 1.9 (0.91) | 2.2 (0.84)
  Week 12 | 1.6 (0.82) | 1.9 (0.93)

7. Secondary Outcome: GAS Score as Evaluated by the Care Giver or the Participant at Week 6 and Week 12
Description: The care giver or participant used the GAS to assess response to treatment at each visit after injection. The assessor was the same throughout the study period. GAS scores were assessed by using the 9-point GAS (-4, -3, -2, -1, -0, +1, +2, +3, +4; -4=very marked worsening, 0=unchanged, +4=very marked improvement) at Week 6 and Week 12.
Time Frame: Week 6 and Week 12
Population: FAS Population. The missing data imputation method was used for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 53 | 53
scores on a scale
  Week 6 | 1.8 (0.91) | 2.1 (0.85)
  Week 12 | 1.6 (0.81) | 1.7 (0.91)

8. Secondary Outcome: Mean Change From Baseline in Red Blood Cell (RBC) Count at the Exit Visit
Description: Blood samples of participants were collected and evaluated for RBC count at Baseline and at the exit visit. Change from Baseline was calculated as the value at the exit visit (Week 12 or earlier) minus the value at Baseline.
Time Frame: Baseline (Day 0) and exit visit (Week 12 or earlier)
Population: Safety Set Population: all enrolled and treated participants. Only those participants for whom data were available for both the Baseline and exit visits were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per Liter
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 47 | 44
10^12 cells per Liter | -0.050 (0.3682) | -0.039 (0.3087)

9. Secondary Outcome: Mean Change From Baseline in White Blood Cell (WBC) and Platelet Count at the Exit Visit
Description: Blood samples of participants were collected and evaluated for WBC count and platelet count at Baseline and at the exit visit. Change from Baseline was calculated as the value at the exit visit (Week 12 or earlier) minus the value at Baseline.
Time Frame: Baseline (Day 0) and the exit visit (Week 12 or earlier)
Population: Safety Set Population. Only those participants for whom data were available for both the Baseline and exit visits were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per Liter
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 47 | 44
10^9 cells per Liter
  WBCs | 0.111 (1.3340) | -0.273 (2.1714)
  Platelets | -10.660 (38.8734) | -1.386 (41.5828)

10. Secondary Outcome: Mean Change From Baseline in the Percentage of Neutrophils, the Percentage of Lymphocytes, the Percentage of Monocytes, the Percentage of Eosinophils, and the Percentage of Basophils at the Exit Visit
Description: Blood samples of participants were collected and evaluated for the percentage of neutrophils, lymphocytes, monocytes, eosinophils, and basophils comprising the total WBC count in the blood at Baseline and at the exit visit. Change from Baseline was calculated as the value at the exit visit (Week 12 or earlier) minus the value at Baseline.
Time Frame: Baseline (Day 0) and the exit visit (Week 12 or earlier)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage of the total WBC
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 47 | 44
Percentage of the total WBC
  Neutrophils | -0.009 (6.3905) | -0.757 (7.8585)
  Lymphocytes | 0.118 (6.4613) | 0.734 (6.7396)
  Monocytes | -0.217 (1.6570) | 0.55 (2.7845)
  Eosinophils | 0.094 (1.3067) | 0.49 (2.3799)
  Basophils | 0.032 (0.2920) | 0.010 (0.2185)

11. Secondary Outcome: Mean Change From Baseline in Hemoglobin Content at the Exit Visit
Description: Blood samples of participants were collected and evaluated for hemoglobin at Baseline and at the exit visit. Change from Baseline was calculated as the value at the exit visit (Week 12 or earlier) minus the value at Baseline.
Time Frame: Baseline (Day 0) and the exit visit (Week 12 or earlier)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Grams per Liter (grams/L)
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 47 | 44
Grams per Liter (grams/L) | -0.255 (10.9989) | -1.409 (8.7559)

12. Secondary Outcome: Mean Change From Baseline in Hematocrit Value at the Exit Visit
Description: The hematocrit, also called packed cell volume or erythrocyte volume fraction, is the volume percentage of red blood cells in the blood. Change from Baseline was calculated as the value at the exit visit (Week 12 or earlier) minus the value at Baseline.
Time Frame: Baseline (Day 0) and the exit visit (Week 12 or earlier)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 47 | 44
percentage | -0.003 (0.0254) | -0.007 (0.0257)

13. Secondary Outcome: Mean Change From Baseline in Total Protein and Albumin Values at the Exit Visit
Description: Blood samples of participants were collected for a biochemical test of total protein and albumin, at Baseline and at the exit visit. Change from Baseline was calculated as the value at the exit visit (Week 12 or earlier) minus the value at Baseline.
Time Frame: Baseline (Day 0) and the exit visit (Week 12 or earlier)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: grams/L
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 47 | 44
grams/L
  Total Protein | -0.711 (5.8908) | -1.484 (6.0077)
  Albumin | -0.400 (3.5067) | -0.236 (4.4753)

14. Secondary Outcome: Mean Change From Baseline in Serum Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Gamma-glutamyl Transferase (y-GT), and Alkaline Phosphatase (ALP) Values at the Exit Visit
Description: Blood samples of participants were collected and evaluated for liver function, including measuring ALT, AST, y-GT, and ALP. Change from Baseline was calculated as the value at the exit visit (Week 12 or earlier) minus the value at Baseline.
Time Frame: Baseline (Day 0) and the exit visit (Week 12 or earlier)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 47 | 44
International Units per Liter (IU/L)
  ALT, n=47, 44 | -1.100 (10.9938) | -0.005 (13.6079)
  AST, n=47, 44 | -0.153 (9.3633) | -0.302 (8.2277)
  y-GT, n=47, 44 | -1.098 (14.0099) | 0.316 (17.4397)
  ALP, n=46, 44 | -3.087 (10.4821) | -4.225 (17.2055)

15. Secondary Outcome: Mean Change From Baseline in Serum Creatinine, Uric Acid, and Total Bilirubin Values at the Exit Visit
Description: Blood samples of participants were collected for a biochemical test of creatine, uric acid, and total bilirubin. Creatine and uric acid are evaluated for kidney function. The liver function test includes total bilirubin. Change from Baseline was calculated as the value at the exit visit (Week 12 or earlier) minus the value at Baseline.
Time Frame: Baseline (Day 0) and the exit visit (Week 12 or earlier)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Micromoles per Liter (μmol/L)
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 47 | 44
Micromoles per Liter (μmol/L)
  Creatinine | -1.509 (9.8783) | -0.984 (20.1303)
  Uric Acid | -3.670 (61.1350) | -16.198 (67.7636)
  Total Bilirubin | 0.249 (4.6873) | -0.293 (3.6399)

16. Secondary Outcome: Mean Change From Baseline in Serum Blood Urea Nitrogen (BUN), Fasting Blood Glucose (FBG), Sodium, Potassium, Chloride, Total Cholesterol, and Triglyceride Values at the Exit Visit
Description: Blood samples of participants were collected for biochemical tests of BUN, FBG, electrolytes, cholesterol, and triglycerides. The BUN test is primarily used to evaluate kidney function. Electrolytes include sodium, potassium, and chloride. Change from Baseline was calculated as the value at the exit visit minus the value at Baseline.
Time Frame: Baseline (Day 0) and the exit visit (Week 12 or earlier)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 47 | 44
Millimoles per Liter (mmol/L)
  BUN, n=47, 44 | -0.292 (1.1855) | 0.226 (2.9929)
  FBG, n=47, 43 | 0.209 (1.3513) | -0.081 (0.8000)
  Sodium, n=47, 44 | 0.423 (3.5990) | -0.034 (2.7857)
  Potassium, n=47, 44 | -0.008 (0.4014) | -0.060 (0.5128)
  Chloride, n=47, 44 | 1.077 (4.0509) | -0.143 (3.4336)
  Total cholesterol, n=47, 43 | -0.057 (0.8410) | 0.282 (0.9535)
  Triglycerides, n=47, 43 | -0.039 (0.6525) | 0.119 (0.5698)

17. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities of Urinalysis at the Screening and Exit Visits
Description: Urine samples of participants were collected for urinalysis, including measuring protein, blood, leukocyte, glucose, and urobilinogen. All values out of the normal range were evaluated by the investigator. Classification of clinically significant and not clinically significant was based on the investigator's clinical judgment; no specific criteria were used.
Time Frame: Screening visit (-Week 1) and the exit visit (Week 12 or earlier)
Population: Safety Set Population. Only those participants for whom data were available for both the Screening and exit visits were analyzed.
Measure: Number; unit: participants
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 47 | 44
participants
  Urine protein, Screening | 0 | 0
  Urine protein, Exit visit | 0 | 0
  Blood, Screening | 0 | 3
  Blood, Exit visit | 0 | 1
  Leukocytes, Screening | 1 | 3
  Leukocytes, Exit visit | 1 | 0
  Urine glucose, Screeing | 2 | 3
  Urine glucose, Exit visit | 0 | 2
  Urobilinogen, Screening | 0 | 0
  Urobilinogen, Exit visit | 0 | 0

18. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (BP) and Diastolic BP at the Exit Visit
Description: Systolic blood pressure (SBP) and diastolic BP of participants were measured in the sitting position. Change from Baseline was calculated as the value at the exit visit (Week 12 or earlier) minus the value at Baseline.
Time Frame: Baseline (Day 0) and the exit visit (Week 12 or earlier)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 47 | 46
Millimeters of mercury (mmHg)
  Systolic BP | -3.1 (8.96) | -2.3 (10.02)
  Diastolic BP | -1.4 (6.27) | -2.5 (7.79)

19. Secondary Outcome: Mean Change From Baseline in Pulse Rate at the Exit Visit
Description: The pulse rate of participants was recorded. Change from Baseline was calculated as the value at the exit visit (Week 12 or earlier) minus the value at Baseline.
Time Frame: Baseline (Screening) and the exit visit (Week 12 or earlier)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Number analyzed (Participants) | 47 | 46
beats per minute | -3.0 (9.27) | 1.0 (8.49)

ADVERSE EVENTS:
Time Frame: Serious and non-serious adverse events were collected from the Screening visit (-1 Week) until the end of study visit (Week 12) or earlier, in case of early withdrawal.
Description: Serious and non-serious adverse events were collected in members of the Safety Set Population, which included all of the enrolled and treated participants.
Arm/Group | BOTOX in Original DB Study; BOTOX in OL Study | Placebo in Original DB Study; BOTOX in OL Study
Serious Adverse Events (participants affected / at risk) | 1/53 | 0/56
Other Adverse Events (participants affected / at risk) | 4/53 | 7/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX in Original DB Study; BOTOX in OL Study (N=53) | Placebo in Original DB Study; BOTOX in OL Study (N=56)
Cerebral arteriovenous malformation haemorrhagic (Congenital, familial and genetic disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX in Original DB Study; BOTOX in OL Study (N=53) | Placebo in Original DB Study; BOTOX in OL Study (N=56)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 3
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Protein total decreased (Investigations) | 0 | 1
Renal function test abnormal (Investigations) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.